CLINICAL TRIAL: NCT03983239
Title: A Phase 1, Open-label, 2-part Study to Evaluate the Effect of Rifampin and Efavirenz on the Pharmacokinetics of Fedratinib in Healthy Adult Subjects
Brief Title: Effect of Rifampin and Efavirenz on the Pharmacokinetics of Fedratinib in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Impact Biomedicines, Inc., a wholly owned subsidiary of Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FEDR-CP-002; U1111-1233-7946 (Other: WHO)
Expanded Access: NCT03723148 (Available)
Record Dates: First submitted 2019-06-03; First posted 2019-06-12 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Subject; Fedratinib; Rifampin; Efavirenz; Drug Interaction
MeSH Terms: interventions — fedratinib; Rifampin; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fedratinib plus Rifampin (Experimental): A single dose of fedratinib on Day 1. On Days 9 through 18, once-daily (QD) doses of rifampin. On Day 17, a single dose of fedratinib will be concomitantly administered with rifampin.
  Interventions: Drug: Fedratinib; Drug: Rifampin; Drug: Efavirenz
- Fedratinib plus Efavirenz (Experimental): A single dose of fedratinib on Day 1. On Days 9 through 18, once-daily (QD) doses of efavirenz. On Day 17, a single dose of fedratinib will be concomitantly administered with efavirenz.
  Interventions: Drug: Fedratinib; Drug: Rifampin; Drug: Efavirenz

INTERVENTIONS:
Drug: Fedratinib — Fedratinib
Drug: Rifampin — Rifampin
Drug: Efavirenz — Efavirenz

SUMMARY:
This is a 2-part study to evaluate the effect of multiple doses of rifampin or efavirenz on the PK, safety, and tolerability of single doses of fedratinib in healthy subjects. Each study part will consist of a nonrandomized, fixed-sequence, open-label design. The study parts can be run in any order or in parallel. Subjects may participate in one part only. For each part, subjects will participate as follows:

* Screening
* Treatment period (includes baseline)
* Follow-up telephone call (4 days [± 2 days] after discharge) During the study, blood samples will be collected at prespecified times for PK. Subject safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject must be willing and able to communicate with the investigator and to adhere to the study visit schedule and other protocol requirements.
3. Subject must be a male or female of any race from ≥ 18 and ≤ 65 years of age at the time of signing the informed Consent Form (ICF).
4. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle-stimulating hormone [FSH] level in the post-menopausal range according to the laboratory used at Screening).
5. Females of childbearing potential (FCBP) must:

   1. Have a negative pregnancy test as verified by the investigator at Screening and Baseline (prior to starting study treatment). She must agree to ongoing pregnancy testing during the course of the study, as applicable, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use, and be able to comply with, any one of the following highly effective contraception methods without interruption, beginning at least 14 days prior to starting investigational product (IP), during the study treatment, and for at least 30 days after the last dose of IP:

      * Intrauterine device (IUD; non-hormonal only); tubal ligation; or a partner with a vasectomy. The chosen form of birth control must be effective by the time the subject receives the first dose of IP.
6. Male subjects must:

   a. Practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made from natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while receiving study treatment, during any dose interruptions, and for at least 30 days after the last dose of IP, even if he has undergone a successful vasectomy.
7. Must have a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
8. Must be healthy, as determined by the investigator on the basis of medical history, physical examination (PE), clinical laboratory test results, vital signs, and 12-lead ECG at screening and check-in (Day -1), as applicable:

   Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin must be at or below the upper limit of the reference range, on or before check-in (Day -1). Other clinical laboratory results must be either within normal range or deemed not clinically significant by the investigator. Any out of range lab tests may be repeated up to one time during the screening period and up to one time at check-in per Investigator discretion to confirm eligibility.
9. Must be afebrile (febrile is defined as ≥ 38°C or 100.3°F).
10. Supine systolic blood pressure (BP) must be in the range of 90 to 140 mmHg (inclusive), supine diastolic BP must be in the range of 50 to 90 mmHg (inclusive), and pulse rate must be in the range of 40 to 100 bpm (inclusive) at screening. Repeat vital signs may be measured at investigator discretion.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening; male subjects must have a corrected QT interval using Fridericia's formula (QTcF) value ≤ 430 msec and females must have a QTcF value ≤ 450 msec. An ECG may be repeated up to two times, and the average of the QTcF values will be used to determine subject eligibility.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. History (ie, within 3 years) of any clinically significant neurological, GI, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other major disorders as determined by the investigator.
2. Any condition, including the presence of laboratory abnormalities, that places the subject at unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable).
3. Subject has prior history of Wernicke's Encephalopathy (WE).
4. Subject has signs or symptoms of WE (eg, severe ataxia, ocular paralysis, or cerebellar signs) without documented exclusion of WE by thiamine level and brain MRI.
5. Subject has thiamine deficiency, defined as thiamine levels in whole blood below normal range according to institutional standard.
6. Subject has active tuberculosis or another disease caused by mycobacteria.
7. Use of any prescribed systemic or topical medication, including vaccines, within 30 days of the first dose administration (with the exception of any odansetron administered for purposes of this study).
8. Use of any nonprescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 14 days of the first dose administration (with the exception of acetaminophen up to 2 grams/day for no more than 3 consecutive days to treat minor illness or headache [per Investigator judgment]).
9. Use of any metabolic enzyme inhibitors or inducers that would affect the relevant drugs within 30 days of the first dose administration unless determined by the investigator that there will be no impact on the study integrity or subject safety. The Indiana University "P450 Drug Interaction Table" should be used to determine inhibitors and/or inducers of metabolic enzymes. The sponsor should be contacted for questions about potential drug-drug interactions and exclusions/prohibitions when necessary.
10. Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
11. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion (eg, bariatric procedure). Appendectomy and cholecystectomy are acceptable.
12. Donated blood or plasma within 8 weeks before the first dose administration.
13. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing or positive drug screening test reflecting consumption of illicit drugs.
14. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing or positive alcohol screen.
15. Known to have serum hepatitis; known to be a carrier of the hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs), hepatitis B core antibody (anti-HBc), or hepatitis C antibody (HCV Ab); have a positive result to the test for hepatitis B or hepatitis C virus at screening or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening. Subjects whose results are compatible with prior immunization (including natural and vaccination) against hepatitis B may be included at the discretion of the investigator.
16. Use of tobacco- or nicotine-containing products within 3 months prior to check-in.
17. Subject has received live vaccination (excluding seasonal flu vaccination) within 90 days of first dosing.
18. History of multiple drug allergies (ie, two or more).
19. Allergic to or hypersensitive to any of the drugs used in the part of the study in which the subject will participate.
20. Has any medical condition, medical history, or use of concomitant medication that is contraindicated in the applicable drug labeling.
21. Female subject who is pregnant or breastfeeding.
22. Subject is part of the clinical staff personnel or a family member of the clinical site staff.
23. Subject has a hypersensitivity to ondansetron.
24. History of severe or serious psychiatric disease ever requiring hospitalization or use of antipsychotic/neuroleptic medications, history of suicidal ideation or suicidal attempt, or undergoing psychiatric treatment will be excluded from study participation.
25. Subject deemed by the investigator or medical professional to be a fall risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Fedratinib Pharmacokinetic - Cmax | Up to approximately 8 days.
  Maximum observed plasma concentration
Fedratinib Pharmacokinetic - Tmax | Up to approximately 8 days.
  Time to maximum observed plasma concentration
Fedratinib Pharmacokinetic - AUC0-t | Up to approximately 8 days.
  Area under the curve from time zero to the last quantifiable concentration
Fedratinib Pharmacokinetic - AUC0-∞ | Up to approximately 8 days.
  Area under the curve from time zero extrapolated to infinity
Fedratinib Pharmacokinetic - t1/2 | Up to approximately 8 days.
  Terminal elimination half-life
Fedratinib Pharmacokinetic - CL/F | Up to approximately 8 days.
  Apparent total plasma clearance when dosed orally
Fedratinib Pharmacokinetic - Vz/F | Up to approximately 8 days.
  Apparent total volume of distribution when dosed orally

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 30 days after completion of study treatment
  Number of participants with an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene
Locations (1):
- Covance Clinical Research Unit Inc - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Ogasawara K, Kam J, Thomas M, Liu L, Liu M, Xue Y, Surapaneni S, Carayannopoulos LN, Zhou S, Palmisano M, Krishna G. Effects of strong and moderate CYP3A4 inducers on the pharmacokinetics of fedratinib in healthy adult participants. Cancer Chemother Pharmacol. 2021 Sep;88(3):369-377. doi: 10.1007/s00280-021-04292-4. Epub 2021 May 21. PMID 34019108